CLINICAL TRIAL: NCT00239343
Title: Randomised Placebo-controlled Phase II Trial of Preoperative Therapy With Gefitinib (Iressa®/ZD1839) and Epirubicin-Cyclophosphamide in Patients With Primary Operable (T2-T3) Oestrogen Receptor Negative Breast Cancer
Brief Title: Phase II Trial of Preoperative Therapy With Gefitinib and Chemotherapy in Patients With ERneg Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0712
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
The aim of the study is to estimate the effect of preoperative gefitinib on the complete pathological response rate in primary estrogen receptor negative breast cancer at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed oestrogen receptor negative primary breast cancer, tumour stage T2-3, N0-2, M0. Eligible for surgery, WHO performance score 0-1.

Exclusion Criteria:

* any prior anticancer therapy including gefitinib (Iressa®), epirubicin (Farmorubicin™), or cyclophosphamide, distant metastases or bilateral breast cancer, any evidence of clinically active interstitial lung disease , other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ, pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
the complete pathological response rate in the two study groups at trial closure

SECONDARY OUTCOMES:
complete and overall objective tumuor response at trial closure according to the RECIST criteria in the per-protocol population

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Director, MD, Study Director — AstraZeneca
Locations (8):
- Denmark (5):
  - Research Site, Århus C
  - Research Stie, Herlev
  - Research Site, København N
  - Research Site, København Ø
  - Research Site, Vejle
- Norway (2):
  - Research Site, Oslo
  - Research Site, Trondheim
- Research Site, Lund, Sweden